CLINICAL TRIAL: NCT00866788
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Dose-Ranging Study of Xolair (Omalizumab) in Patients With Chronic Idiopathic Urticaria (CIU) Who Remain Symptomatic With Antihistamine Treatment (H1)
Brief Title: A Study of Xolair (Omalizumab) in Patients With Chronic Idiopathic Urticaria (CIU) Who Remain Symptomatic With Antihistamine Treatment (H1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Q4577g
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2011-09-09 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Chronic Idiopathic Urticaria
Keywords: Xolair; CIU
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Omalizumab 75 mg (Experimental): Omalizumab (Xolair) was administered subcutaneously on Day 0 of the study. Participants remained on stable doses of their pre-allocation Chronic Idiopathic Urticaria (CIU) H1 antihistamine treatment throughout the study, and were provided diphenhydramine as rescue medication for pruritus relief on an as-needed basis.).
  Interventions: Drug: omalizumab; Drug: H1 antihistamines; Drug: Diphenhydramine
- Omalizumab 300 mg (Experimental): Omalizumab (Xolair) was administered subcutaneously on Day 0 of the study. Participants remained on stable doses of their pre-allocation Chronic Idiopathic Urticaria (CIU) H1 antihistamine treatment throughout the study, and were provided diphenhydramine as rescue medication for pruritus relief on an as-needed basis.
  Interventions: Drug: omalizumab; Drug: H1 antihistamines; Drug: Diphenhydramine
- Omalizumab 600 mg (Experimental): Omalizumab (Xolair) was administered subcutaneously on Day 0 of the study. Participants remained on stable doses of their pre-allocation Chronic Idiopathic Urticaria (CIU) H1 antihistamine treatment throughout the study, and were provided diphenhydramine as rescue medication for pruritus relief on an as-needed basis.
  Interventions: Drug: omalizumab; Drug: H1 antihistamines; Drug: Diphenhydramine
- Placebo (Placebo Comparator): Participants received a single subcutaneous placebo injection on Day 0 of the study. Participants remained on stable doses of their pre-allocation Chronic Idiopathic Urticaria CIU) H1 antihistamine treatment throughout the study, and were provided diphenhydramine as rescue medication for pruritus relief on an as-needed basis.
  Interventions: Drug: omalizumab; Drug: placebo; Drug: H1 antihistamines; Drug: Diphenhydramine

INTERVENTIONS:
Drug: omalizumab — Administered by subcutaneous injection
  Other Names: Xolair
Drug: placebo — Participants received a single subcutaneous placebo injection on Day 0 of the study.
  Arms: Placebo
Drug: H1 antihistamines — Patients received one of the following: Cetirizine 10 mg once per day (QD), Levocetirizine dihydrochloride 5 mg QD, Fexofenadine 60 mg twice per day or 180 mg QD, Loratadine 10 mg QD or Desloratadine 5 mg QD
Drug: Diphenhydramine — Diphenhydramine was provided and used on an as-needed basis (25 mg per dose)

SUMMARY:
The study is a Phase II, dose-ranging, multicenter, randomized, double-blind, placebo-controlled, parallel-group study of the efficacy and safety of a single subcutaneously administered omalizumab dose as add-on therapy for the treatment of adolescent and adult patients 12-75 years old who have been diagnosed with CIU and remain symptomatic despite treatment with therapeutic doses of an H1 antihistamine. The study will enroll approximately 76 patients at approximately 45 study centers in the United States and Germany.

ELIGIBILITY:
Inclusion Criteria:

* CIU diagnosis > 3 months (by history)
* No underlying etiology clearly defined for urticaria (main manifestation cannot be physical urticaria)

Exclusion Criteria:

* Pregnant, breastfeeding, or women not taking contraception
* Patients < 40kg
* Treatment with any investigational agent within 30 days of screening
* Recent history of drug or alcohol abuse
* Atopic dermatitis or other skin disease associated with pruritus
* Clinically relevant major systemic disease (making interpretation of the study results difficult)
* Previously treated with omalizumab (< 12 months since last injection)
* Patients may not take during treatment period or have been taking within the past 3 months any of the following medications/treatments: regular (daily/every other day) hydroxychloroquine, methotrexate, cyclosporine, cyclophosphamide, IVIG, or plasmapheresis
* Patients may not have been taking doxepin within the past 6 weeks regular (daily/every other day).

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Rosen, M.D., Ph.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab 75 mg; Omalizumab 600 mg: Omalizumab (Xolair) was administered subcutaneously on Day 0 of the study. Participants remained on stable doses of their pre-allocation Chronic Idiopathic Urticaria (CIU) H1 antihistamine treatment throughout the study, and were provided diphenhydramine as rescue medication for pruritus relief on an as-needed basis.
- Omalizumab 300 mg: Omalizumab (Xolair) was administered subcutaneously on Day 0 of the study. Participants remained on stable doses of their pre-allocation Chronic Idiopathic Urticaria (CIU)H1 antihistamine treatment throughout the study, and were provided diphenhydramine as rescue medication for pruritus relief on an as-needed basis.
Period: Overall Study
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Started | 21 | 23 | 25 | 21
Completed | 15 | 17 | 23 | 16
Not Completed | 6 | 6 | 2 | 5
Not completed — Adverse Event | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Disease progression | 3 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg | Total
Number analyzed (Participants) | 21 | 23 | 25 | 21 | 90
Age, Customized [Number; unit: participants]
  12-<18 years | 2 | 2 | 1 | 0 | 5
  18-<40 years | 7 | 10 | 12 | 11 | 40
  >=40 years | 12 | 11 | 12 | 10 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 17 | 12 | 61
  Male | 4 | 8 | 8 | 9 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Urticaria Activity Score 7 (UAS7) From Baseline to Week 4
Description: The UAS is a composite diary-recorded score, which is the sum of the numeric severity intensity ratings (0 = none to 3 = intense) for 1) the number of wheals (hives) and 2) the intensity of the pruritus (itch). The UAS7 is the sum of the daily average UAS (morning and evening values) for 7 days. The maximum UAS7 score is 42.
Time Frame: Baseline (based on the 7 days prior to randomization) and 4 weeks (Days 21-27)
Population: Intent-to-Treat population (all randomized patients). The last observation carried forward value was used if a patient's Week 4 diary data were completely missing. One subject from the omalizumab 600-mg group did not have any post-baseline data and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Number analyzed (Participants) | 21 | 23 | 25 | 20
scores on a scale | -6.91 (9.84) | -9.79 (11.75) | -19.93 (12.38) | -14.56 (10.17)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; Test type: Superiority or Other; p = 0.1601, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 300 mg; Test type: Superiority or Other; p = 0.0003, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 600 mg; Test type: Superiority or Other; p = 0.0473, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)

2. Secondary Outcome: Change in the Weekly Pruritus Score From Baseline to Week 4
Description: The pruritus (itch) score was recorded by participants twice daily (morning and evening) based on the severity of itch over the last 12 hours, using a scale from 0 (none) to 3 (severe). The weekly pruritus score was the sum of average daily pruritus scores over the previous 7 days. The range of the weekly score is 0-21.
Time Frame: Baseline (based on the 7 days prior to randomization) and 4 weeks (Days 21-27)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Number analyzed (Participants) | 21 | 23 | 25 | 20
scores on a scale | -3.45 (5.22) | -4.50 (5.84) | -9.22 (5.98) | -6.46 (5.63)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; Test type: Superiority or Other; p = 0.1640, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 300 mg; Test type: Superiority or Other; p = 0.0005, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 600 mg; Test type: Superiority or Other; p = 0.0558, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)

3. Secondary Outcome: Change in the Weekly Score for Number of Hives From Baseline to Week 4
Description: The number of hives was recorded by participants twice daily (morning and evening) using a scale from 0 (no hives) to 3 (more than 12 hives). The weekly score of number of hives was the sum of the average daily scores over the previous 7 days, and ranged from 0 to 21.
Time Frame: Baseline (based on the 7 days prior to randomization) and 4 weeks (Days 21-27)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Number analyzed (Participants) | 21 | 23 | 25 | 20
scores on a scale | -3.46 (5.17) | -5.28 (6.91) | -10.71 (6.75) | -8.10 (6.00)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; Test type: Superiority or Other; p = 0.1411, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 300 mg; Test type: Superiority or Other; p = 0.0003, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 600 mg; Test type: Superiority or Other; p = 0.0248, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)

4. Secondary Outcome: Change in the Weekly Score for Sleep Interference From Baseline to Week 4
Description: The extent to which hives or itch interfered with participants' sleep was recorded once daily in the patient diary using a scale from 0 (no interference) to 3 (substantial interference, waking often). The weekly score of sleep interference was the sum of the daily scores over the previous 7 days, and ranged from 0 to 21.
Time Frame: Baseline (based on the 7 days prior to randomization) and 4 weeks (Days 21-27)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Number analyzed (Participants) | 21 | 23 | 25 | 20
scores on a scale | -3.23 (5.93) | -3.90 (5.03) | -5.81 (5.36) | -6.85 (6.23)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; Test type: Superiority or Other; p = 0.5507, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 300 mg; Test type: Superiority or Other; p = 0.1525, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 600 mg; Test type: Superiority or Other; p = 0.0449, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)

5. Secondary Outcome: Change in the Weekly Score for the Amount of Rescue Medication From Baseline to Week 4
Description: Diphenhydramine 25mg was provided and used on an as-needed basis (maximum 3 times/day) as rescue medication. The weekly score for the amount of rescue medication is the sum of the daily scores for the amount of rescue medication used at each day in the week, and ranged from 0 to 21.
Time Frame: Baseline (based on the 7 days prior to randomization) and 4 weeks (Days 21-27)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Pills
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Number analyzed (Participants) | 21 | 23 | 25 | 20
Pills | -1.38 (4.39) | -1.74 (4.48) | -2.64 (5.17) | -1.69 (3.56)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; Test type: Superiority or Other; p = 0.7261, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 300 mg; Test type: Superiority or Other; p = 0.162, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 600 mg; Test type: Superiority or Other; p = 0.6504, van Elteren test — The p-value was based on the van Elteren test (stratified by baseline weight ≥ 80 or < 80 kg)

6. Secondary Outcome: Number of Patients With Adverse Events by Severity
Description: The severity (i.e. intensity) of each Adverse Event (AE) was graded according to the following scale: Mild: Symptoms causing no or minimal interference with usual social and functional activities. Moderate: Symptoms causing greater than minimal interference with usual social and functional activities. Severe: Symptoms causing inability to perform usual social and functional activities.
  Additional AE data is provided in the AE section below. The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an AE. A "Serious" AE is defined below.
Time Frame: 16 weeks overall (data reported separately for "up to 4 weeks" and "Weeks 5 to 16")
Population: Safety-Evaluable Population, which included all randomized patients who received any study drug. number (n) equals (=) number of participants analyzed in the specified category.
Measure: Number; unit: participants
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Number analyzed (Participants) | 21 | 23 | 25 | 21
participants
  4 Weeks - Any Adverse Event (n=21,23,25,21) | 10 | 8 | 12 | 10
  4 Weeks - Mild (n=21,23,25,21) | 8 | 4 | 6 | 7
  4 Weeks - Moderate (n=21,23,25,21) | 2 | 3 | 5 | 2
  4 Weeks - Severe (n=21,23,25,21) | 0 | 1 | 1 | 1
  Follow-up period-Any adverse event (n=20,18,23,20) | 7 | 9 | 12 | 5
  Follow-up period-Mild (n=20,18,23,20) | 4 | 5 | 4 | 3
  Follow-up period-Moderate (n=20,18,23,20) | 2 | 2 | 6 | 1
  Follow-up period-Severe (n=20,18,23,20) | 1 | 2 | 2 | 1

7. Secondary Outcome: Number of Participants With Immunogenicity
Description: Immunogenicity was measured by detection of anti-therapeutic antibodies (anti-omalizumab antibodies) using a fragment enzyme-linked immunosorbent assay (ELISA).
Time Frame: 16 weeks
Population: Safety-Evaluable Population
Measure: Number; unit: participants
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Number analyzed (Participants) | 21 | 23 | 25 | 21
participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Maximum Observed Concentration (Cmax) of Omalizumab
Description: Cmax is the maximum (or peak) concentration of omalizumab in serum.
Time Frame: Pre-dose and 2 hours post-dose on Days 0 and 3 of Week 0, Weeks 1, 2, 3, 4, 8, 12, 16 or early termination (up to Week 16)
Population: Pharmacokinetic-Evaluable Population included all randomized participants who received omalizumab and had pharmacokinetic data available. Here, number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Number analyzed (Participants) | 22 | 23 | 20
micrograms per milliliter (µg/mL) | 11.4 (16.4) | 33.1 (10.4) | 67 (26.9)

9. Secondary Outcome: Time to Maximum Concentration (Tmax) of Omalizumab
Description: Tmax is the time to maximum concentration of omalizumab.
Time Frame: as for outcome 8
Population: Pharmacokinetic-Evaluable Population; Here, number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Number analyzed (Participants) | 22 | 23 | 20
days | 7.37 (3.72) | 8.01 (5.54) | 6.24 (3.51)

10. Secondary Outcome: Area Under the Concentration-time Curve From Time of Dosing Extrapolated to Infinity (AUC-Inf)
Description: AUCinf is the area under the concentration-time curve from time of dosing extrapolated to infinity. AUCinf was measured in microgram times day per milliliter (µg*day/mL). Only participants having complete profiles and completed the study were included in the analysis.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: µg*day/mL
Arm/Group | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Number analyzed (Participants) | 18 | 22 | 19
µg*day/mL | 317 (99.6) | 1260 (580) | 2800 (1140)

11. Secondary Outcome: Terminal Half-Life (t1/2) of Omalizumab
Description: Terminal Half-Life (t1/2) is the time required for the serum concentration of omalizumab to decrease by half in the final stage of its elimination.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Number analyzed (Participants) | 18 | 22 | 19
days | 18.2 (4.76) | 17.1 (4.41) | 22.5 (5.9)

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from Day -7 until end of study at 16 weeks.
Description: A Serious AE is any AE that is either:
  * Fatal
  * Life threatening
  * Requires or prolongs inpatient hospitalization
  * Results in persistent or significant disability/incapacity
  * A congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the study treatment
  * Considered a significant medical event by the investigator
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 300 mg | Omalizumab 600 mg
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23 | 1/25 | 0/21
Other Adverse Events (participants affected / at risk) | 5/21 | 9/23 | 11/25 | 8/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Omalizumab 75 mg (N=23) | Omalizumab 300 mg (N=25) | Omalizumab 600 mg (N=21)
Chest Pain (General disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Omalizumab 75 mg (N=23) | Omalizumab 300 mg (N=25) | Omalizumab 600 mg (N=21)
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 3 | 2
Nasopharyngitis (Infections and infestations) | 1 | 4 | 3 | 1
Headache (Nervous system disorders) | 1 | 0 | 2 | 3
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Idiopathic Uticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights."